CLINICAL TRIAL: NCT05012215
Title: Ultrasound Guided Thoracic Paravertebral Block Versus Ultrasound Guided Caudal Epidural Block in Pediatric Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Paravertebral Versus Caudal Block in Pediatric PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Paravertebral Caudal PCNL
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Kidney Stones; Percutaneous Nephrolithotomy
Keywords: paravertebral block; caudal block; Percutaneous nephrolithotomy; pediatric
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paravertebral (Experimental): Ultrasound-guided thoracic paravertebral block
  Interventions: Procedure: Paravertebral
- Caudal (Active Comparator): Caudal block
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Paravertebral — Ultrasound-guided paravertebral block
  Arms: Paravertebral
Procedure: Caudal block — Caudal block
  Arms: Caudal

SUMMARY:
To compare the efficacy of Ultrasound guided thoracic paravertebral block versus ultrasound guided caudal epidural block in pediatric patients undergoing percutaneous nephrolithotomy

DETAILED DESCRIPTION:
Percutaneous Nephrolithotomy (PCNL) is a commonly performed surgical procedure for complex upper renal tract calculi. Although the skin incision for PCNL appears small, the intensity of intraoperative and postoperative pain is significant owing to soft tissue injury.

Paravertebral block is the technique of injecting local anesthetics in a space immediately lateral to where the spinal nerves emerge from the intervertebral foramina. This technique is used increasingly for intra-operative and post-operative.

Caudal epidural block involves placing a needle through the sacral hiatus to deliver medications into the epidural space. This approach is used widely used for surgical anesthesia and analgesia in pediatric patients.

this work aims to compare the efficacy of Ultrasound guided thoracic paravertebral block versus ultrasound guided caudal epidural block in pediatric patients undergoing percutaneous nephrolithotomy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous nephrolithotomy

Exclusion Criteria:

* Coagulation disorders
* Infection at the site of injection
* Allergy to the local anesthetics used
* Spinal cord abnormalities or neurological deficits

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Blood pressure during surgery in mmHg | through the surgery, an average of 2 hours
Heart rate (beats/minute) | through the surgery, an average of 2 hours
The concentration of sevoflurane in % | through the surgery, an average of 2 hours
Postoperative pain using FLACC score | up to 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt